CLINICAL TRIAL: NCT02253043
Title: The Safety and Efficacy of Long-term Treatment of PINS Stimulator System for Patients With Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-002
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): DBS Implant and stimulation
  Interventions: Device: Deep Brain Stimulation (Beijing PINS Medical Co., Ltd)

INTERVENTIONS:
Device: Deep Brain Stimulation (Beijing PINS Medical Co., Ltd) — PINS Stimulator System
  Other Names: Deep Brain Stimulation Device

SUMMARY:
Purpose: The purpose of this clinical study is to verify the long term effectiveness and safety of a bilateral deep brain stimulation (DBS) produced by Beijing PINS Medical Co., Ltd. as a treatment option for patients with cognitive, behavioral, and functional disability of Alzheimer's disease.

DETAILED DESCRIPTION:
Other: Deep Brain Stimulation Implanted device Subjects will then be instructed to apply PINS Deep Brain Stimulation Device for 12 month.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 40 to 80 years old;
2. Subject with AD diagnosed according to the criteria for probable AD as defined by the National Institute of Neurological Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA);
3. Subject have received the diagnosis of AD within the past 2 years;
4. Subject have a CDR of 0.5 or 1.0;
5. Score between 20 and 28 on the Mini Mental State Examination
6. have been taking a stable dose of cholinesterase inhibitors for a minimum of 6 months.

Exclusion Criteria:

1. Patients with hearing impairment;
2. Failures of important organs and in severe conditions
3. Be reluctant or disabled to receive neuropsychological assessments;
4. Participate in other clinical trial;
5. Has a life expectancy of < 1 year.
6. The investigator and/or enrollment review committee, would preclude participation in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-Cog) | 12 month
  Change from Baseline

SECONDARY OUTCOMES:
Clinical Dementia Rating Scale | 12 month
  Change from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - 301 Hospatl, Beijing, Beijing Municipality